CLINICAL TRIAL: NCT02631525
Title: A Comparison of Post-operative Recovery Between Remifentanil-propofol and Remifentanil-desflurane Anesthesia Guided by Bispectral Index Monitoring
Brief Title: Recovery Profile Comparison Between Remifentanil-propofol or Desflurane Anesthesia Monitored With Bispectral Index.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Baxter Healthcare Corporation (Industry); Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Renato Santiago Gomez, Head of surgery department of the Medical School of the Federal University of Minas Gerais, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE - 31820014.8.0000.5149
Record Dates: First submitted 2015-12-04; First posted 2015-12-16 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Delayed Emergence From Anesthesia
Keywords: Airway extubation; Anesthesia Recovery Period; Desflurane; Propofol; Intravenous anesthesia; Balanced Anesthesia
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- REM-PRO (Active Comparator): Total intravenous anesthesia with remifentanil and propofol, target controlled infusion based on Minto's and Marsh's pharmacokinetic models.
  Interventions: Drug: Propofol
- REM-DES (Active Comparator): Balanced anesthesia with remifentanil target controlled infusion based on Minto's pharmacokinetic model and desflurane.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Desflurane — Balanced anesthesia with remifentanil and desflurane guided by bispectral monitoring
  Arms: REM-DES
Drug: Propofol — Total intravenous anesthesia based on propofol
  Other Names: Diprivan
  Arms: REM-PRO

SUMMARY:
Bispectral monitoring anesthesia with remifentanil-desflurane has a better post-operative recovery than remifentanil-propofol.

DETAILED DESCRIPTION:
It is a randomized, double blind study, involving 40 adult female patients submitted to general anesthesia. The patients were distributed into 2 groups: remifentanil-propofol-based anesthesia and remifentanil-desflurane-based anesthesia groups. Bispectral index (BIS) monitoring guided the anesthesia by setting target BIS range value between 40 and 60. Anesthetics were adjusted to reached that. Primary outcome was: extubation time (time from anesthetic discontinuation to endotracheal tube cuff). Secondary measured outcomes: intra-operative cardiovascular drug use; time to follow command before extubation; protective airway reflex recovery time after extubation. Protective airway reflex test recovery was performed at predetermined time intervals (2, 6, 14, 22 and 30 minutes) from the time to follow a standard command until the first demonstrated ability to swallow 20 ml of water in an upright position.Post-anesthesia care unit recovery data were also recorded: Ramsay sedation scale; vital signs, post-operative pain; morphine consumption.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over 18 years old classified by the American Society of Anesthesiologists as physical status I or II, undergoing elective breast surgery with general anesthesia.

Exclusion Criteria:

* History of: illegal drug and alcohol abuse
* Pregnancy on course or suspicion of
* Neuromuscular disorders
* Cerebral vascular disease
* Dysphagia
* Dysphonia
* Gastroesophageal reflux disease
* Previous larynx and/or upper gastrointestinal tract surgery
* Allergy to any drug to be used and malignant hyperthermia.
* Patients who develop hemodynamic instability in the surgery and need blood transfusion were excluded from the study.
* Patients unable to swallow 20 ml of water in an upright position were also excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato S Gomez, PhD, Principal Investigator — Professor of the Medicine School of the Federal University of Minas Gerais

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu ZF, Jian GS, Lee MS, Lin C, Chen YF, Chen YW, Huang YS, Cherng CH, Lu CH. An analysis of anesthesia-controlled operating room time after propofol-based total intravenous anesthesia compared with desflurane anesthesia in ophthalmic surgery: a retrospective study. Anesth Analg. 2014 Dec;119(6):1393-406. doi: 10.1213/ANE.0000000000000435. PMID 25211391
- [Background] Mckay RE, Large MJC, Balea MC, Mckay WR. Airway reflexes return more rapidly after desflurane anesthesia than after sevoflurane anesthesia. Anesth Analg. 2005 Mar;100(3):697-700. doi: 10.1213/01.ANE.0000146514.65070.AE. PMID 15728054
- [Background] Wachtel RE, Dexter F, Epstein RH, Ledolter J. Meta-analysis of desflurane and propofol average times and variability in times to extubation and following commands. Can J Anaesth. 2011 Aug;58(8):714-24. doi: 10.1007/s12630-011-9519-1. Epub 2011 Jun 1. PMID 21630118
- [Background] Punjasawadwong Y, Phongchiewboon A, Bunchungmongkol N. Bispectral index for improving anaesthetic delivery and postoperative recovery. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD003843. doi: 10.1002/14651858.CD003843.pub3. PMID 24937564

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | REM-PRO | REM-DES
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REM-PRO | REM-DES | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (15) | 46 (11) | 50 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Extubation Time
Description: Time from anesthetic discontinuation to endotracheal tube cuff deflation
Time Frame: Time from anesthetic discontinuation to endotracheal tube cuff deflation
Measure: Mean (Full Range); unit: minutes
Arm/Group | REM-PRO | REM-DES
Number analyzed (Participants) | 19 | 20
minutes | 9.5 [4.9 to 14.4] | 6.2 [3.1 to 18.5]

ADVERSE EVENTS:
Arm/Group | REM-PRO | REM-DES
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No